CLINICAL TRIAL: NCT00581581
Title: Long-term Follow-up After Head Cooling for Neonatal Encephalopathy
Brief Title: CoolCap Followup Study-Coordination of Participating Centers
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: Olympic Medical (Industry)
Responsible Party: Principal Investigator, Ronnie Guillet, Professor, University of Rochester
Other Study IDs: RSRB00020479
Record Dates: First submitted 2007-12-21; First posted 2007-12-27 (Estimated); Results first posted 2013-03-08 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Neonatal Encephalopathy
Keywords: neonatal encephalopathy; therapeutic hypothermia; head cooling; neonatal asphyxia
MeSH Terms: conditions — Asphyxia Neonatorum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Randomized to cooling (original randomized clinical trial): All children, now 6-8 years old who were randomized to cooling in the original trial were included in this arm. Cooling was achieved via the CoolCap system (Olympic Medical/Natus Corporation) in these babies.
- 2: Randomized to standard care (original randomized clinical trial): All children, now 6-8 years old, who were treated using the standard of care at the time (normal temperature) were included in this arm. Infants' temperatures were monitored per standard of care. Most infants were cared for on an open wamer that was servo-controlled to normal body temperature (37 C) or in a standard bassinette.

SUMMARY:
This observational study will assess long-term functional outcome of survivors from neonatal encephalopathy who were previously treated with either head cooling or with conventional care in a randomized clinical trial. Children's parents will be interviewed by phone by trained staff using the WeeFIM questionnaire to ascertain the childrens' functional performance on a set of skills basic to daily life. This instrument is able to assess a very wide range of abilities, from independently functioning to needing total assistance. The ratings will be used to examine the relationship between the outcome previously measured at 18 months age and functional outcome at school age and to triage the children into those who clearly could not be tested on standardized exams of cognitive functioning, those who potentially could, even if at a low level of cognitive ability, and those who appear to be functioning at an age-appropriate level.

DETAILED DESCRIPTION:
Previous studies have demonstrated that hypothermia for hypoxic-ischemic encephalopathy in the neonatal period is generally safe and feasible, and can improve intermediate term survival without handicap. There is, however, no information on whether cooling improves longer term (school-age) outcomes in non-handicapped survivors. The current observational trial is designed to help obtain additional followup information on children who participated in the initial randomized clinical trial of head-cooling for neonatal encephalopathy. A first step is to collect information on the current status (at 7-8 years of age) of participants in the original study using a standardized telephone questionnaire. This will allow the investigators to more appropriately target children for whom further, more detailed, in-person neurodevelopmental testing would be appropriate. Given limited resources, identification of children for whom such testing would be helpful and instructive is a necessary goal.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in the CoolCap study
* Survivors to 7-8 years of age
* Parental consent to participation

Exclusion Criteria:

* Lack of parental consent

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Eligible children will be those who participated in the original randomized clinical trial, "Brain Cooling for the Treatment of Perinatal Hypoxic-Ischemic Encephalopathy". Infants enrolled in that study were randomized to cooling or standard care. Survivors to 7-8 years of age are eligible for this observational followup study.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2007-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Guillet, MD, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Background] Gluckman PD, Wyatt JS, Azzopardi D, Ballard R, Edwards AD, Ferriero DM, Polin RA, Robertson CM, Thoresen M, Whitelaw A, Gunn AJ. Selective head cooling with mild systemic hypothermia after neonatal encephalopathy: multicentre randomised trial. Lancet. 2005 Feb 19-25;365(9460):663-70. doi: 10.1016/S0140-6736(05)17946-X. PMID 15721471
- [Result] Guillet R, Edwards AD, Thoresen M, Ferriero DM, Gluckman PD, Whitelaw A, Gunn AJ; CoolCap Trial Group. Seven- to eight-year follow-up of the CoolCap trial of head cooling for neonatal encephalopathy. Pediatr Res. 2012 Feb;71(2):205-9. doi: 10.1038/pr.2011.30. Epub 2011 Dec 21. PMID 22258133

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals who participated in the parent study (CoolCap) were invited to participate in this follow-up study when they were 7-8 years old. Site investigators contacted prior participants' families by phone for consent. Contact information for the families who consented was provided to a central examiner.
Pre-assignment Details: Observational study - determination of outcome at 7-8 years after prior randomization in parent study to therapeutic hypothermia vs standard of care for infants with hypoxic-ischemic encephalopathy who met eligibility requirements.
Groups:
- Therapeutic Hypothermia: Randomized to cooling (original RCT)
- Standard Care: Randomized to standard care (original RCT)
Period: Overall Study
Arm/Group | Therapeutic Hypothermia | Standard Care
Started | 32 | 30
Completed | 32 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Therapeutic Hypothermia | Standard Care | Total
Number analyzed (Participants) | 32 | 30 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32 | 30 | 62
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 7.68 (0.62) | 7.66 (0.63) | 7.67 (0.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 18 | 30
  Male | 20 | 12 | 32
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 5 | 11
  United States | 24 | 23 | 47
  New Zealand | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: WeeFIM Score
Description: WeeFIM instrument (the Functional Independence Measure for Children, Uniform Data System for Medical Rehabilitation, Buffalo, NY) is a set of ratings of 18 skills divided into 3 general domains: 8 Self-care; 5 Mobility; 5 Cognition. Caregivers rate a child about extent of independence, full functioning, in carrying out each of those 18 skills, on a scale from "1" for total assistance, total dependence, maximal prompting, or not testable to "7" for complete independence. The ratings are combined to yield 3 Domain scores and a WeeFIM Total. Favorable=mean+/-2SD. We are reporting the percentage of participants with a favorable response.
Time Frame: 7-8 years after initial intervention
Measure: Number; unit: percentage of participants
Arm/Group | Therapeutic Hypothermia | Standard Care
Number analyzed (Participants) | 32 | 30
percentage of participants | 78 | 80

ADVERSE EVENTS:
Description: No adverse events were measured; study limited to administration of questionnaire describing function at 7-8 years of age.
Arm/Group | Therapeutic Hypothermia | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No